CLINICAL TRIAL: NCT00622375
Title: A Phase I, Single- And Multiple-Dose, Relative Bioavailability and Pharmacokinetic Study of Encapsulated Mesalamine Granules Administered Orally to Healthy Volunteers
Brief Title: PK Study of Encapsulated Mesalamine Granules in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MPPK1003
Record Dates: First submitted 2008-02-14; First posted 2008-02-25 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Healthy
Keywords: Pharmacokinetic study; Healthy subjects
MeSH Terms: interventions — Mesalamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: mesalamine

INTERVENTIONS:
Drug: mesalamine — encapsulated mesalamine granules

SUMMARY:
The current study is being conducted to evaluate the relative bioavailability and single- and multiple-dose pharmacokinetics of encapsulated mesalamine granules(eMG) in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* The subject is Male, or female of Non-childbearing potentia.l
* The subject is female of childbearing potential, who has a negative serum pregnancy test at screen and agrees to using appropriate birth control.
* The subject is between the ages of 18 and 45 years.
* The subject has a body mass index (BMI) between 18 and 32 kg/m2 (weight/[height]).

Exclusion Criteria:

* The subject is seropositive for human immunodeficiency virus (HIV),hepatitis B surface antigen, and/or hepatitis C virus.
* The subject has any clinically significant medical, social, or emotional problem.
* The subject is pregnant or lactating
* The subject has a history of clinically significant renal, hepatic,endocrine, oncological,gastrointestinal, or cardiovascular disease or a history of epilepsy, asthma, diabetes mellitus, psychosis, glaucoma, or severe head injury.
* The subject is currently receiving mesalamine or aspirin containing products
* The subject has a history of viral, bacterial, or fungal infection within 4 weeks of screening.
* The subject has an acute illness within 1 week of study-drug administration.
* The subject has an abnormal nutritional status, including unconventional, alternative,and abnormal diets; excessive or unusual vitamin intake; malabsorption; psychological eating disorders; difficulty swallowing medication; significant recent weight change; etc.
* The subject has clinically significant allergies.
* The subject has a hypersensitivity or allergy to mesalamine or other salicylate.
* The subject has known or suspected alcohol abuse or illicit drug use within the past year
* The subject has used tobacco (or nicotine products) during the 6 months prior to screening
* The subject has participated in an investigational drug study within the 30 days before receiving study drug

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-02; Primary Completion 2008-02 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Individual pharmacokinetic parameters for mesalamine and its metabolites will be summarized with descriptive statistics | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Shaw, PhD, Study Director — Bausch Health Americas, Inc.
Locations (1):
- Dallas, Texas, United States